CLINICAL TRIAL: NCT05197894
Title: Virtual Reality for Improving Symptoms in Palliative Care
Acronym: VRPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Patricia Valcke, Adjunct Professor, Specialist Palliative Care Consultant, Western University, Schulich School of Medicine and Dentistry, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Windsor Essex Hospice VR
Record Dates: First submitted 2021-11-19; First posted 2022-01-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Cancer and Non-cancer Hospice Patients
Keywords: virtual reality; palliative care; Edmonton symptom assessment scale; Hospice; depression; anxiety; pain; shortness of breath; well-being
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders; Pain; Dyspnea

STUDY DESIGN:
Intervention Model Description: ESAS scores for 5 key symptoms (pain, shortness of breath, depression, anxiety, and well-being) and qualitative question(s) will be asked verbally by one of the investigators and recorded on an ipad directly into the Qualtrics form, before and after the VR session. Vital signs (blood pressure, heart rate, respiratory rate) will also be measured before and after the VR session. Participants will be given a list of VR applications to choose from. They will then be given instructions by a research assistant (approximately 10 minutes) on how to use the selected application using Oculus Quest 2 they have chosen, as well as time for any questions they may have before starting their VR experience. They will then have an approximately 30-minute session of that VR experience. They may or may not be accompanied by a family member or significant other and will also have a research assistant available to aid them in any difficulties experienced during the VR experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR experience (Experimental): Participants will be given a list of VR applications to choose from. They will then be given instructions by a research assistant (approximately 10 minutes) on how to use the selected application they have chosen, as well as time for any questions they may have before starting their VR experience. They will then have an approximately 30-minute session of that VR experience. They may or may not be accompanied by a family member or significant other and will also have a research assistant available to aid them in any difficulties experienced during the VR experience.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — The intervention is a Virtual Reality experience within a selected application using an Oculus Quest 2 ©, as previously in the relevant intervention arm.

SUMMARY:
The objective of this study is to determine whether VR can ameliorate symptoms for palliative care patients within a hospice setting. We also aim to verify the efficacy with a larger sample size than previously shown, as well as extend the population to include non-cancer patients receiving Hospice care. We will further attempt to delineate whether there is a sustainability of symptomatic improvement one week after VR experiences.

DETAILED DESCRIPTION:
Potential candidates will be provided with our assent and consent information form and the study will be explained to them in detail prior to gaining consent. As per standard practice at The Hospice of Windsor & Essex County, palliative care ESAS symptoms will be measured at baseline during the week prior to the VR experience. The mean of these pre-VR scores will be calculated as a baseline, optimally 3 separate ESAS scores in the preceding week. ESAS symptoms and expectations/satisfaction will then be measured immediately before and after the VR experience. An average set of ESAS scores will then be calculated in the same manner for one week post VR as per baseline pre-VR scores above.

We expect to find a decrease in Palliative Care symptoms after the intervention of a VR experience.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years or older
* admitted to Hospice for Specialty Palliative Care

Exclusion Criteria:

* Palliative Performance Scale (PPS) ≤ 20%
* severe cognitive impairment leading to inability to provide ESAS scores for 5 key symptoms measured in this study
* severe visual and/or hearing impairment preventing use of VR (glasses and hearing aids may be worn during VR sessions and do not exclude participation)
* absolute inability to sit
* paralysis of an upper limb
* participant dies before VR experience

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
VR experience effect on pain, shortness of breath, depression, anxiety, and well-being scores (0 - 10) | ESAS scores measured immediately before VR experience will be compared to ESAS scores measured immediately after VR experience
  The primary outcome of this study will be a significant difference in change of ESAS score for 5 key symptoms (pain, shortness of breath, depression, anxiety, and well-being) immediately before and after a VR experience.

SECONDARY OUTCOMES:
VR experience longitudinal effect (one week later) on baseline pain, shortness of breath, depression, anxiety, and well-being scores (0 - 10) | Baseline average ESAS scores measured one week prior to the VR experience will be compared to the average of ESAS scores one week following the VR experience.
  The first secondary outcome of this study will be a significant difference between the mean of the 1-week pre-VR and the mean of the 1-week post-VR ESAS scores for 5 key symptoms (pain, shortness of breath, depression, anxiety, and well-being). For more objective evaluation of pain and distress we will also be measuring vitals immediately before and immediately after each VR experience.
VR experience effect on Mean Arterial Pressure (MAP) (part of vital signs) as indicator for Pain and/or Distress | MAP measured immediately before and immediately after each VR experience.
  For more objective evaluation of pain and distress, the investigators will be measuring blood pressure to compare the Mean Arterial Pressure (MAP; mmHg) immediately before and immediately after each VR experience.
VR experience effect on Heart Rate (HR) (part of vital signs) as indicator for Pain and/or Distress | HR measured immediately before and immediately after each VR experience.
  For more objective evaluation of pain and distress, the investigators will be measuring Heart Rate (HR; beats per minute [bpm]) immediately before and immediately after each VR experience.
VR experience effect on Respiratory Rate (RR) (part of vital signs) as indicator for Pain and/or Distress | RR measured immediately before and immediately after each VR experience.
  For more objective evaluation of pain and distress, the investigators will be measuring Respiratory Rate (RR; breaths per minute [brpm]) immediately before and immediately after each VR experience.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospice of Windsor and Essex County, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to make individual participant data (IPD) available to other researchers.